CLINICAL TRIAL: NCT05105542
Title: Muscarinic M1 Receptor Availability and Cognition in Schizophrenia
Brief Title: M1 Schizophrenia PET Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rajiv Radhakrishnan, MD, Assistant Professor of Psychiatry, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000031171; 1R21MH123870-01A1 (NIH); 1R01MH113557-01 (NIH)
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Healthy
Keywords: Schizophrenia; Muscarinic M1 Receptor; M1 AChR; [11C]EMO; PET Scan; MRI Scan
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Receptor, Muscarinic M1; Positron-Emission Tomography

STUDY DESIGN:
Intervention Model Description: Two groups will be studied: 1.) patients diagnosed with schizophrenia or schizoaffective disorder, and 2.) age and gender-matched healthy controls. Both groups will undergo neuroimaging, cognitive assessments, etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Schizophrenia or schizoaffective disorder (Experimental): Participants will undergo a single PET scan with [11C]EMO ≤ 20 mCi
  Interventions: Drug: 11C-EMO - A Novel PET Radiotracer for Muscarinic M1 Receptor; Device: PET Scan
- Healthy Controls (Experimental): Participants will undergo a single PET scan with [11C]EMO ≤ 20 mCi
  Interventions: Drug: 11C-EMO - A Novel PET Radiotracer for Muscarinic M1 Receptor; Device: PET Scan

INTERVENTIONS:
Drug: 11C-EMO - A Novel PET Radiotracer for Muscarinic M1 Receptor — The radiotracer, [11C]EMO, will be administered at the beginning of each PET scan.
Device: PET Scan — PET scanner with high sensitivity and resolution available for human brain imaging

SUMMARY:
This exploratory study seeks to examine M1 receptor availability in SZ patients and to relate M1 receptor availability to proximal and distal measures of cognitive performance, namely evoked ɣ oscillations in the EEG and verbal memory. Furthermore, the relationship between hippocampal [11C]EMO availability (BPND), evoked ɣ oscillations, verbal memory, and measures of illness severity will be explored.

DETAILED DESCRIPTION:
Converging lines of evidence from postmortem studies provide strong evidence that brain muscarinic M1 receptor deficit is present in a subset of schizophrenia (SZ) patients. M1 receptors are an important target for cognitive deficits in SZ. However, until now, it has not been possible to examine the heterogeneity of SZ with respect to M1 receptor availability in vivo. The development of a novel positron emission tomography (PET) ligand, [11C]EMO, at Yale PET Center provides a unique opportunity to, for the first time, examine in vivo brain muscarinic M1 receptor availability in SZ and, concurrently, elucidate the relationship of M1 receptors to cognitive deficits in SZ.

The investigators will compare M1 receptor availability in SZ patients and age-, gender-matched healthy controls using [11C]EMO and the High Resolution Research Tomograph (HRRT), a PET scanner with high sensitivity and resolution available for human brain imaging. This study will explore the relationship between: hippocampal [11C]EMO binding (as a measure of hippocampal M1 AChR availability), encoding-related γ power during a verbal memory task, verbal memory, gender, and serum acetylcholine level. This exploratory study will provide the necessary pilot data to conduct a larger study to fully investigate the heterogeneity of SZ with respect to M1 receptor availability.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18- 65 years that are physically and mentally healthy with the exception of DSM-5 schizophrenia or schizoaffective disorder diagnosis
* Subjects with no metal in the body that may pose a risk during MRI scanning
* No significant medical history, including head trauma and bleeding disorders

Exclusion Criteria:

* Men and women with a history or presence of clinically significant medical conditions
* People who suffer from claustrophobia, have MRI incompatible implants, or other contraindications for MRI and PET scans

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Hippocampal M1 availability | 10 days
  Measured by [11C]EMO availability (BPND)

SECONDARY OUTCOMES:
evoked ɣ oscillations | 10 days
  Measured by EEG
verbal memory | 10 days
  Measured by cognitive assessments

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Radhakrishnan, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mogg AJ, Eessalu T, Johnson M, Wright R, Sanger HE, Xiao H, Crabtree MG, Smith A, Colvin EM, Schober D, Gehlert D, Jesudason C, Goldsmith PJ, Johnson MP, Felder CC, Barth VN, Broad LM. In Vitro Pharmacological Characterization and In Vivo Validation of LSN3172176 a Novel M1 Selective Muscarinic Receptor Agonist Tracer Molecule for Positron Emission Tomography. J Pharmacol Exp Ther. 2018 Jun;365(3):602-613. doi: 10.1124/jpet.117.246454. Epub 2018 Apr 11. PMID 29643252
- [Background] Oki T, Takagi Y, Inagaki S, Taketo MM, Manabe T, Matsui M, Yamada S. Quantitative analysis of binding parameters of [3H]N-methylscopolamine in central nervous system of muscarinic acetylcholine receptor knockout mice. Brain Res Mol Brain Res. 2005 Jan 5;133(1):6-11. doi: 10.1016/j.molbrainres.2004.09.012. PMID 15661360
- [Background] Smart K, Gallezot JD, Nabulsi N, Labaree D, Zheng MQ, Huang Y, Carson RE, Hillmer AT, Worhunsky PD. Separating dopamine D2 and D3 receptor sources of [11C]-(+)-PHNO binding potential: Independent component analysis of competitive binding. Neuroimage. 2020 Jul 1;214:116762. doi: 10.1016/j.neuroimage.2020.116762. Epub 2020 Mar 19. PMID 32201327
- [Background] Worhunsky PD, Matuskey D, Gallezot JD, Gaiser EC, Nabulsi N, Angarita GA, Calhoun VD, Malison RT, Potenza MN, Carson RE. Regional and source-based patterns of [11C]-(+)-PHNO binding potential reveal concurrent alterations in dopamine D2 and D3 receptor availability in cocaine-use disorder. Neuroimage. 2017 Mar 1;148:343-351. doi: 10.1016/j.neuroimage.2017.01.045. Epub 2017 Jan 19. PMID 28110088
- [Background] Carruthers SP, Van Rheenen TE, Gurvich C, Sumner PJ, Rossell SL. Characterising the structure of cognitive heterogeneity in schizophrenia spectrum disorders. A systematic review and narrative synthesis. Neurosci Biobehav Rev. 2019 Dec;107:252-278. doi: 10.1016/j.neubiorev.2019.09.006. Epub 2019 Sep 7. PMID 31505202
- [Background] Niendam TA, Ray KL, Iosif AM, Lesh TA, Ashby SR, Patel PK, Smucny J, Ferrer E, Solomon M, Ragland JD, Carter CS. Association of Age at Onset and Longitudinal Course of Prefrontal Function in Youth With Schizophrenia. JAMA Psychiatry. 2018 Dec 1;75(12):1252-1260. doi: 10.1001/jamapsychiatry.2018.2538. PMID 30285056
- [Background] Van Rheenen TE, Cropley V, Zalesky A, Bousman C, Wells R, Bruggemann J, Sundram S, Weinberg D, Lenroot RK, Pereira A, Shannon Weickert C, Weickert TW, Pantelis C. Widespread Volumetric Reductions in Schizophrenia and Schizoaffective Patients Displaying Compromised Cognitive Abilities. Schizophr Bull. 2018 Apr 6;44(3):560-574. doi: 10.1093/schbul/sbx109. PMID 28981831
- [Background] Wells R, Swaminathan V, Sundram S, Weinberg D, Bruggemann J, Jacomb I, Cropley V, Lenroot R, Pereira AM, Zalesky A, Bousman C, Pantelis C, Weickert CS, Weickert TW. The impact of premorbid and current intellect in schizophrenia: cognitive, symptom, and functional outcomes. NPJ Schizophr. 2015 Nov 4;1:15043. doi: 10.1038/npjschz.2015.43. eCollection 2015. PMID 27336046
- [Background] Scarr E, Craig JM, Cairns MJ, Seo MS, Galati JC, Beveridge NJ, Gibbons A, Juzva S, Weinrich B, Parkinson-Bates M, Carroll AP, Saffery R, Dean B. Decreased cortical muscarinic M1 receptors in schizophrenia are associated with changes in gene promoter methylation, mRNA and gene targeting microRNA. Transl Psychiatry. 2013 Feb 19;3(2):e230. doi: 10.1038/tp.2013.3. PMID 23423139
- [Background] Scarr E, Hopper S, Vos V, Seo MS, Everall IP, Aumann TD, Chana G, Dean B. Low levels of muscarinic M1 receptor-positive neurons in cortical layers III and V in Brodmann areas 9 and 17 from individuals with schizophrenia. J Psychiatry Neurosci. 2018 Aug;43(5):338-346. doi: 10.1503/jpn.170202. PMID 30125244
- [Background] Hopper S, Pavey GM, Gogos A, Dean B. Widespread Changes in Positive Allosteric Modulation of the Muscarinic M1 Receptor in Some Participants With Schizophrenia. Int J Neuropsychopharmacol. 2019 Oct 1;22(10):640-650. doi: 10.1093/ijnp/pyz045. PMID 31428788
- [Background] Crook JM, Tomaskovic-Crook E, Copolov DL, Dean B. Decreased muscarinic receptor binding in subjects with schizophrenia: a study of the human hippocampal formation. Biol Psychiatry. 2000 Sep 1;48(5):381-8. doi: 10.1016/s0006-3223(00)00918-5. PMID 10978721
- [Background] Lebois EP, Trimper JB, Hu C, Levey AI, Manns JR. Effects of Selective M1 Muscarinic Receptor Activation on Hippocampal Spatial Representations and Neuronal Oscillations. ACS Chem Neurosci. 2016 Oct 19;7(10):1393-1405. doi: 10.1021/acschemneuro.6b00160. Epub 2016 Aug 12. PMID 27479319
- [Background] Harrison PJ. Using our brains: the findings, flaws, and future of postmortem studies of psychiatric disorders. Biol Psychiatry. 2011 Jan 15;69(2):102-3. doi: 10.1016/j.biopsych.2010.09.008. No abstract available. PMID 21183008
- [Background] Nabulsi NB, Holden D, Zheng MQ, Bois F, Lin SF, Najafzadeh S, Gao H, Ropchan J, Lara-Jaime T, Labaree D, Shirali A, Slieker L, Jesudason C, Barth V, Navarro A, Kant N, Carson RE, Huang Y. Evaluation of 11C-LSN3172176 as a Novel PET Tracer for Imaging M1 Muscarinic Acetylcholine Receptors in Nonhuman Primates. J Nucl Med. 2019 Aug;60(8):1147-1153. doi: 10.2967/jnumed.118.222034. Epub 2019 Feb 7. PMID 30733324
- [Background] Green MF, Kern RS, Heaton RK. Longitudinal studies of cognition and functional outcome in schizophrenia: implications for MATRICS. Schizophr Res. 2004 Dec 15;72(1):41-51. doi: 10.1016/j.schres.2004.09.009. PMID 15531406
- [Background] Barch DM, Ceaser A. Cognition in schizophrenia: core psychological and neural mechanisms. Trends Cogn Sci. 2012 Jan;16(1):27-34. doi: 10.1016/j.tics.2011.11.015. Epub 2011 Dec 12. PMID 22169777
- [Background] Green MF, Harvey PD. Cognition in schizophrenia: Past, present, and future. Schizophr Res Cogn. 2014 Mar;1(1):e1-e9. doi: 10.1016/j.scog.2014.02.001. PMID 25254156
- [Background] Carruthers SP, Gurvich CT, Rossell SL. The muscarinic system, cognition and schizophrenia. Neurosci Biobehav Rev. 2015 Aug;55:393-402. doi: 10.1016/j.neubiorev.2015.05.011. Epub 2015 May 21. PMID 26003527
- [Background] Marino MJ, Rouse ST, Levey AI, Potter LT, Conn PJ. Activation of the genetically defined m1 muscarinic receptor potentiates N-methyl-D-aspartate (NMDA) receptor currents in hippocampal pyramidal cells. Proc Natl Acad Sci U S A. 1998 Sep 15;95(19):11465-70. doi: 10.1073/pnas.95.19.11465. PMID 9736760
- [Background] Levey AI, Kitt CA, Simonds WF, Price DL, Brann MR. Identification and localization of muscarinic acetylcholine receptor proteins in brain with subtype-specific antibodies. J Neurosci. 1991 Oct;11(10):3218-26. doi: 10.1523/JNEUROSCI.11-10-03218.1991. PMID 1941081
- [Background] Anagnostaras SG, Murphy GG, Hamilton SE, Mitchell SL, Rahnama NP, Nathanson NM, Silva AJ. Selective cognitive dysfunction in acetylcholine M1 muscarinic receptor mutant mice. Nat Neurosci. 2003 Jan;6(1):51-8. doi: 10.1038/nn992. PMID 12483218
- [Background] Gould RW, Dencker D, Grannan M, Bubser M, Zhan X, Wess J, Xiang Z, Locuson C, Lindsley CW, Conn PJ, Jones CK. Role for the M1 Muscarinic Acetylcholine Receptor in Top-Down Cognitive Processing Using a Touchscreen Visual Discrimination Task in Mice. ACS Chem Neurosci. 2015 Oct 21;6(10):1683-95. doi: 10.1021/acschemneuro.5b00123. Epub 2015 Aug 5. PMID 26176846
- [Background] Cropley VL, Scarr E, Fornito A, Klauser P, Bousman CA, Scott R, Cairns MJ, Tooney PA, Pantelis C, Dean B. The effect of a muscarinic receptor 1 gene variant on grey matter volume in schizophrenia. Psychiatry Res. 2015 Nov 30;234(2):182-7. doi: 10.1016/j.pscychresns.2015.09.004. Epub 2015 Sep 10. PMID 26481978
- [Background] Liao DL, Hong CJ, Chen HM, Chen YE, Lee SM, Chang CY, Chen H, Tsai SJ. Association of muscarinic m1 receptor genetic polymorphisms with psychiatric symptoms and cognitive function in schizophrenic patients. Neuropsychobiology. 2003;48(2):72-6. doi: 10.1159/000072880. PMID 14504414
- [Background] Scarr E, Cowie TF, Kanellakis S, Sundram S, Pantelis C, Dean B. Decreased cortical muscarinic receptors define a subgroup of subjects with schizophrenia. Mol Psychiatry. 2009 Nov;14(11):1017-23. doi: 10.1038/mp.2008.28. Epub 2008 Mar 4. PMID 18317461
- [Background] Green MF, Horan WP, Lee J. Nonsocial and social cognition in schizophrenia: current evidence and future directions. World Psychiatry. 2019 Jun;18(2):146-161. doi: 10.1002/wps.20624. PMID 31059632
- [Background] Mesholam-Gately RI, Giuliano AJ, Goff KP, Faraone SV, Seidman LJ. Neurocognition in first-episode schizophrenia: a meta-analytic review. Neuropsychology. 2009 May;23(3):315-36. doi: 10.1037/a0014708. PMID 19413446
- [Background] Arnedo J, Svrakic DM, Del Val C, Romero-Zaliz R, Hernandez-Cuervo H; Molecular Genetics of Schizophrenia Consortium; Fanous AH, Pato MT, Pato CN, de Erausquin GA, Cloninger CR, Zwir I. Uncovering the hidden risk architecture of the schizophrenias: confirmation in three independent genome-wide association studies. Am J Psychiatry. 2015 Feb 1;172(2):139-53. doi: 10.1176/appi.ajp.2014.14040435. Epub 2014 Oct 31. PMID 25219520
- [Background] Bakker G, Vingerhoets C, Boucherie D, Caan M, Bloemen O, Eersels J, Booij J, van Amelsvoort T. Relationship between muscarinic M1 receptor binding and cognition in medication-free subjects with psychosis. Neuroimage Clin. 2018 Mar 3;18:713-719. doi: 10.1016/j.nicl.2018.02.030. eCollection 2018. PMID 29560312
- [Background] Lavalaye J, Booij J, Linszen DH, Reneman L, van Royen EA. Higher occupancy of muscarinic receptors by olanzapine than risperidone in patients with schizophrenia. A[123I]-IDEX SPECT study. Psychopharmacology (Berl). 2001 Jun;156(1):53-7. doi: 10.1007/s002130000679. PMID 11465633
- [Background] Raedler TJ. Comparison of the in-vivo muscarinic cholinergic receptor availability in patients treated with clozapine and olanzapine. Int J Neuropsychopharmacol. 2007 Apr;10(2):275-80. doi: 10.1017/S1461145706006584. Epub 2006 Apr 6. PMID 16945161
- [Background] Erskine D, Taylor JP, Bakker G, Brown AJH, Tasker T, Nathan PJ. Cholinergic muscarinic M1 and M4 receptors as therapeutic targets for cognitive, behavioural, and psychological symptoms in psychiatric and neurological disorders. Drug Discov Today. 2019 Dec;24(12):2307-2314. doi: 10.1016/j.drudis.2019.08.009. Epub 2019 Sep 6. PMID 31499186
- [Background] Nathan PJ, Watson J, Lund J, Davies CH, Peters G, Dodds CM, Swirski B, Lawrence P, Bentley GD, O'Neill BV, Robertson J, Watson S, Jones GA, Maruff P, Croft RJ, Laruelle M, Bullmore ET. The potent M1 receptor allosteric agonist GSK1034702 improves episodic memory in humans in the nicotine abstinence model of cognitive dysfunction. Int J Neuropsychopharmacol. 2013 May;16(4):721-31. doi: 10.1017/S1461145712000752. Epub 2012 Aug 29. PMID 22932339
- [Background] Shekhar A, Potter WZ, Lightfoot J, Lienemann J, Dube S, Mallinckrodt C, Bymaster FP, McKinzie DL, Felder CC. Selective muscarinic receptor agonist xanomeline as a novel treatment approach for schizophrenia. Am J Psychiatry. 2008 Aug;165(8):1033-9. doi: 10.1176/appi.ajp.2008.06091591. Epub 2008 Jul 1. PMID 18593778
- [Background] Han M, Newell K, Zavitsanou K, Deng C, Huang XF. Effects of antipsychotic medication on muscarinic M1 receptor mRNA expression in the rat brain. J Neurosci Res. 2008 Feb 1;86(2):457-64. doi: 10.1002/jnr.21491. PMID 17787019
- [Background] Carson RE, Barker WC, Liow J-S, Adler S, Johnson CA. Design of a motion-compensation OSEM List-mode Algorithm for Resolution-Recovery Reconstruction of the HRRT. IEEE Nuclear Science Symposium and Medical Imaging Conference; 2003; Portland, OR; 2003. p. M16-6.
- [Background] Jin X, Mulnix T, Sandiego CM, Carson RE. Evaluation of frame-based and event-by-event motion-correction methods for awake monkey brain PET imaging. J Nucl Med. 2014 Feb;55(2):287-93. doi: 10.2967/jnumed.113.123299. Epub 2014 Jan 16. PMID 24434295
- [Background] Horti AG, Fan H, Kuwabara H, Hilton J, Ravert HT, Holt DP, Alexander M, Kumar A, Rahmim A, Scheffel U, Wong DF, Dannals RF. 11C-JHU75528: a radiotracer for PET imaging of CB1 cannabinoid receptors. J Nucl Med. 2006 Oct;47(10):1689-96. PMID 17015906
- [Background] Gallezot JD, Nabulsi N, Neumeister A, Planeta-Wilson B, Williams WA, Singhal T, Kim S, Maguire RP, McCarthy T, Frost JJ, Huang Y, Ding YS, Carson RE. Kinetic modeling of the serotonin 5-HT(1B) receptor radioligand [(11)C]P943 in humans. J Cereb Blood Flow Metab. 2010 Jan;30(1):196-210. doi: 10.1038/jcbfm.2009.195. Epub 2009 Sep 23. PMID 19773803
- [Background] Tzourio-Mazoyer N, Landeau B, Papathanassiou D, Crivello F, Etard O, Delcroix N, Mazoyer B, Joliot M. Automated anatomical labeling of activations in SPM using a macroscopic anatomical parcellation of the MNI MRI single-subject brain. Neuroimage. 2002 Jan;15(1):273-89. doi: 10.1006/nimg.2001.0978. PMID 11771995
- [Background] Innis RB, Cunningham VJ, Delforge J, Fujita M, Gjedde A, Gunn RN, Holden J, Houle S, Huang SC, Ichise M, Iida H, Ito H, Kimura Y, Koeppe RA, Knudsen GM, Knuuti J, Lammertsma AA, Laruelle M, Logan J, Maguire RP, Mintun MA, Morris ED, Parsey R, Price JC, Slifstein M, Sossi V, Suhara T, Votaw JR, Wong DF, Carson RE. Consensus nomenclature for in vivo imaging of reversibly binding radioligands. J Cereb Blood Flow Metab. 2007 Sep;27(9):1533-9. doi: 10.1038/sj.jcbfm.9600493. Epub 2007 May 9. PMID 17519979
- [Background] Lammertsma AA, Hume SP. Simplified reference tissue model for PET receptor studies. Neuroimage. 1996 Dec;4(3 Pt 1):153-8. doi: 10.1006/nimg.1996.0066. PMID 9345505
- [Background] Wu Y, Carson RE. Noise reduction in the simplified reference tissue model for neuroreceptor functional imaging. J Cereb Blood Flow Metab. 2002 Dec;22(12):1440-52. doi: 10.1097/01.WCB.0000033967.83623.34. PMID 12468889
- [Background] Babiloni C, Vecchio F, Mirabella G, Buttiglione M, Sebastiano F, Picardi A, Di Gennaro G, Quarato PP, Grammaldo LG, Buffo P, Esposito V, Manfredi M, Cantore G, Eusebi F. Hippocampal, amygdala, and neocortical synchronization of theta rhythms is related to an immediate recall during rey auditory verbal learning test. Hum Brain Mapp. 2009 Jul;30(7):2077-89. doi: 10.1002/hbm.20648. PMID 18819109
- [Background] Kay SR, Opler LA, Lindenmayer JP. The Positive and Negative Syndrome Scale (PANSS): rationale and standardisation. Br J Psychiatry Suppl. 1989 Nov;(7):59-67. No abstract available. PMID 2619982
- [Background] Cassetta BD, Menon M, Carrion PB, Pearce H, DeGraaf A, Leonova O, White RF, Stowe RM, Honer WG, Woodward TS, Torres IJ. Preliminary examination of the validity of the NIH toolbox cognition battery in treatment-resistant psychosis. Clin Neuropsychol. 2020 Jul;34(5):981-1003. doi: 10.1080/13854046.2019.1694072. Epub 2019 Nov 29. PMID 31782350
- [Background] Gershon RC, Cella D, Fox NA, Havlik RJ, Hendrie HC, Wagster MV. Assessment of neurological and behavioural function: the NIH Toolbox. Lancet Neurol. 2010 Feb;9(2):138-9. doi: 10.1016/S1474-4422(09)70335-7. No abstract available. PMID 20129161
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Gershon RC, Wagster MV, Hendrie HC, Fox NA, Cook KF, Nowinski CJ. NIH toolbox for assessment of neurological and behavioral function. Neurology. 2013 Mar 12;80(11 Suppl 3):S2-6. doi: 10.1212/WNL.0b013e3182872e5f. PMID 23479538
- [Background] Boozalis T, Teixeira AL, Cho RY, Okusaga O. C-Reactive Protein Correlates with Negative Symptoms in Patients with Schizophrenia. Front Public Health. 2018 Jan 22;5:360. doi: 10.3389/fpubh.2017.00360. eCollection 2017. PMID 29404313
- [Background] Deng H, Kahlon RS, Mohite S, Amin PA, Zunta-Soares G, Colpo GD, Stertz L, Fries GR, Walss-Bass C, Soares JC, Okusaga OO. Elevated Plasma S100B, Psychotic Symptoms, and Cognition in Schizophrenia. Psychiatr Q. 2018 Mar;89(1):53-60. doi: 10.1007/s11126-017-9514-y. PMID 28435992
- [Background] Mohite S, Yang F, Amin PA, Zunta-Soares G, Colpo GD, Stertz L, Sharma AN, Fries GR, Walss-Bass C, Soares JC, Okusaga OO. Plasma soluble L-selectin in medicated patients with schizophrenia and healthy controls. PLoS One. 2017 Mar 23;12(3):e0174073. doi: 10.1371/journal.pone.0174073. eCollection 2017. PMID 28334045
- [Background] Yohn SE, Conn PJ. Positive allosteric modulation of M1 and M4 muscarinic receptors as potential therapeutic treatments for schizophrenia. Neuropharmacology. 2018 Jul 1;136(Pt C):438-448. doi: 10.1016/j.neuropharm.2017.09.012. Epub 2017 Sep 9. PMID 28893562
- [Background] Ranganathan M, Cortes-Briones J, Radhakrishnan R, Thurnauer H, Planeta B, Skosnik P, Gao H, Labaree D, Neumeister A, Pittman B, Surti T, Huang Y, Carson RE, D'Souza DC. Reduced Brain Cannabinoid Receptor Availability in Schizophrenia. Biol Psychiatry. 2016 Jun 15;79(12):997-1005. doi: 10.1016/j.biopsych.2015.08.021. Epub 2015 Aug 29. PMID 26432420
- [Background] D'Souza DC, Esterlis I, Carbuto M, Krasenics M, Seibyl J, Bois F, Pittman B, Ranganathan M, Cosgrove K, Staley J. Lower ss2*-nicotinic acetylcholine receptor availability in smokers with schizophrenia. Am J Psychiatry. 2012 Mar;169(3):326-34. doi: 10.1176/appi.ajp.2011.11020189. PMID 22193533
- [Background] Esterlis I, Ranganathan M, Bois F, Pittman B, Picciotto MR, Shearer L, Anticevic A, Carlson J, Niciu MJ, Cosgrove KP, D'Souza DC. In vivo evidence for beta2 nicotinic acetylcholine receptor subunit upregulation in smokers as compared with nonsmokers with schizophrenia. Biol Psychiatry. 2014 Sep 15;76(6):495-502. doi: 10.1016/j.biopsych.2013.11.001. Epub 2013 Nov 13. PMID 24360979
- [Background] D'Souza DC, Perry E, MacDougall L, Ammerman Y, Cooper T, Wu YT, Braley G, Gueorguieva R, Krystal JH. The psychotomimetic effects of intravenous delta-9-tetrahydrocannabinol in healthy individuals: implications for psychosis. Neuropsychopharmacology. 2004 Aug;29(8):1558-72. doi: 10.1038/sj.npp.1300496. PMID 15173844